CLINICAL TRIAL: NCT03759587
Title: A Phase 2, Multicenter, Open-label, Single-arm Study to Evaluate the Safety of Niraparib in Japanese Patients With Platinum-sensitive, Relapsed Ovarian, Fallopian Tube, or Primary Peritoneal Cancer Who Achieved CR or PR in the Last Chemotherapy Containing Platinum-based Anticancer Agents
Brief Title: Japan Phase 2 Study of Niraparib (Maintenance Therapy) in Participants With Relapsed Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Niraparib-2001; U1111-1222-4074 (Other: WHO); JapicCTI-184225 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2018-11-29; First posted 2018-11-30 (Actual); Results first posted 2020-03-25 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-05

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Niraparib 300 mg (Experimental): Niraparib 300 mg, capsules, orally, once daily on Days 1 to 28 of each 28-day treatment cycle (up to 51 cycles).
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Niraparib capsule

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of niraparib in Japanese participants with platinum-sensitive, relapsed ovarian cancer, fallopian tube cancer, or primary peritoneal cancer who achieved complete response (CR) or partial response (PR) in the last chemotherapy containing platinum-based anticancer agents.

DETAILED DESCRIPTION:
The drug being tested in this study is called niraparib. Niraparib is being tested to treat people who have platinum-sensitive, relapsed ovarian cancer, fallopian tube cancer, or primary peritoneal cancer. This study will look at the safety and efficacy of niraparib in Japanese participants.

The study will enroll approximately 15 participants. Participants will be enrolled to one group and after that will be asked to take niraparib capsules at the same time each day throughout the study:

- Niraparib 300 mg

This multi-center trial will be conducted in Japan. The overall time to participate in this study is approximately 28 months. Participants will make multiple visits to the clinic in the treatment period, and the post-treatment period including follow-up assessments after the last dose of the study drug.

ELIGIBILITY:
Inclusion Criteria

1. Japanese female participants aged 20 years or older on the day of signing informed consent.
2. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.
3. Participant must have a histologically diagnosed ovarian cancer, fallopian tube cancer, or primary peritoneal cancer.
4. Participant must have a high-grade (or Grade 3) serous or high-grade predominantly serous histology or known to have germline breast cancer gene mutation (gBRCAmut).
5. Participants must have completed at least 2 previous lines of platinum-containing therapy (eg, carboplatin, oxaliplatin, or cisplatin):

   Note: The last platinum regimen did not necessarily have to immediately follow the next-to-last (penultimate) platinum regimen. For example, if a participant received a non-platinum regimen between the penultimate platinum regimen and last platinum regimen, she could have been eligible as long as she met all entry criteria.
   1. For the penultimate platinum-based chemotherapy prior to study enrollment, participants must have had platinum-sensitive disease after this treatment, defined as achieving a response (CR or PR) and disease progression >6 months after completion of her last dose of platinum therapy (documented 6 to 12 months or >12 months). Source documentation was required.
   2. For the last line of platinum-based chemotherapy prior to study enrollment:

      * Participants must have received a platinum-containing regimen for a minimum of 4 cycles.
      * Participants must have achieved a partial or complete tumor response.
      * Following the last regimen, participants must have had either: CA-125 in the normal range, OR; CA-125 decrease by more than 90% during the last platinum regimen, and which was stable for at least 7 days (ie, no increase >15%).
      * Following the last regimen, participants could not have had any measurable lesion >2 cm at the time of study enrollment.
   3. Participants must have been enrolled within 8 weeks after completion of their final dose of the platinum-containing regimen.
6. Participants must have performance status of ≤1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status Scale.
7. Participants must have adequate organ function as indicated by the following laboratory values:

   1. Absolute neutrophil count (ANC) ≥1,500/μL.
   2. Platelet count ≥100,000/μL.
   3. Hemoglobin ≥9 g/dL.
   4. Serum creatinine ≤1.5× institutional upper limit of normal (ULN) OR calculated creatinine clearance ≥50 mL/minute, using the Cockcroft-Gault equation.
   5. Total bilirubin ≤1.5×ULN OR direct bilirubin ≤1×ULN.
   6. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN unless liver metastases were present, in which case they had to be ≤5×ULN.
8. Participants must be able to take oral medications.
9. Female participants of childbearing potential must be negative for pregnancy test (beta-human chorionic gonadotropin [β-hCG]) within 7 days prior to receiving the first dose of study treatment.
10. Female participants who:

    1. Are postmenopausal for at least 1 year before the screening visit, OR
    2. Are surgically sterile, OR
    3. If they are of childbearing potential, agree to practice 1 highly effective method of contraception and 1 additional effective (barrier) method at the same time, from the time of signing the informed consent through 180 days after the last dose of study drug, OR
    4. Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods], condoms only, withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.)

Exclusion Criteria

1. Participants who have had drainage of ascites during last 2 cycles of last chemotherapy.
2. Participants who have had palliative radiotherapy encompassing >20% of the bone marrow within 1 week of the first dose of study treatment.
3. Participants who have any, persistent, Grade ≥3 toxicity from last cancer therapy.
4. Participants who have symptomatic, uncontrolled brain or leptomeningeal metastases. To be considered "controlled," central nervous system (CNS) disease must have undergone treatment (eg, radiation or chemotherapy) at least 1 month prior to study enrollment. The participant must not have had any new or progressive signs or symptoms related to the CNS disease and must have been taking a stable dose of steroids or no steroids (as long as these were started at least 4 weeks prior to enrollment] or no steroids). A scan to confirm the absence of brain metastases at baseline was not required. Participants with spinal cord compression might have been considered if they had received definitive treatment for this and evidence of clinically stable disease for 28 days.
5. Participants who have known hypersensitivity to the components of niraparib.
6. Participants who have had prior treatment with a known poly (adenosine diphosphate [ADP]-ribose) polymerase (PARP) inhibitor.
7. Participant who have had treatment with any investigational products within 28 days or 5 half-lives (whichever was longer) before the first dose.
8. Participants who have had major surgery per Investigator judgment within 3 weeks of the first dose. Participant must have recovered from any effects of any major surgery.
9. Participants who have diagnosis, detection, or treatment of invasive second primary malignancy other than ovarian cancer ≤24 months prior to study enrollment (except basal or squamous cell carcinoma of the skin that was definitively treated). Note: Participants must not have any known history or current diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML), irrespective of the time for disease history.
10. Participants who are considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days of the first dose) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, small bowel obstruction or other serious gastrointestinal disorder, or any psychiatric disorder that prohibits obtaining informed consent.
11. Participants who have received a transfusion (platelets or red blood cells) within 4 weeks of the first dose of study treatment.
12. Participants who have received a live virus or bacterial vaccines within 4 weeks of the first dose of study treatment.
13. Participants who have a history or current evidence of any condition, therapy, or lab abnormality (including active or uncontrolled myelosuppression [ie, anemia, leukopenia, neutropenia, thrombocytopenia]) that might confound the results of the study, interfere with the participant's participation throughout the study period, or study participation is not in the best interest of the participant.
14. Participants who are regular user (including "recreational use") of any illicit drugs at the time of signing informed consent or have a recent history (within the past year) of drug or alcohol abuse.
15. Participants who are pregnant or breast-feeding, or expecting to conceive within the planned duration of the study.

    NOTE: If a breast-feeding woman discontinue breast-feeding, she may be enrolled in the study.
16. Participants who are immunocompromised (participants with splenectomy are allowed).
17. Participants who have known human immunodeficiency virus (HIV) positive.
18. Participants who have known hepatitis B surface antigen (HBsAg) positive, or known or suspected active hepatitis C virus (HCV) infection.

NOTE: Participants who are positive for hepatitis B core antibody (HBcAb) or hepatitis B surface antibody (HBsAb) can be enrolled but must have an undetectable hepatitis B virus (HBV) viral load. Participants who have positive hepatitis C virus antibody (HCVAb) must have an undetectable HCV viral load.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female participants with platinum-sensitive, relapsed ovarian cancer, fallopian tube cancer, or primary peritoneal cancer were eligible to be enrolled in this study.
Enrollment: 19 (Actual)
Dates: Start 2018-12-28 (Actual); Primary Completion 2019-03-17 (Actual); Study Completion 2022-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (27):
- Japan (27):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Hirosaki University Hospital, Hirosaki, Aomori
  - Shikoku Cancer Center, Matsuyama, Ehime
  - Ehime University Hospital, Tōon, Ehime
  - Kurume University Hospital, Kurume, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Kansai Rosai Hospital, Amagasaki, Hyōgo
  - Iwate Medical University Hospital, Morioka, Iwate
  - Tokai University Hospital, Isehara, Kanagawa
  - Nippon Medical School Musashi Kosugi Hospital, Kawasaki, Kanagawa
  - Mie University Hospital, Tsu, Mie-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - University of the Ryukyus Hospital, Nakagami-gun, Okinawa
  - Kindai University Hospital, Sayama, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Shizuoka Cancer Center, Nagaizumi-cho, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Cancer Institute Hospital, Koto-ku, Tokyo
  - The Jikei University Hospital, Minato-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Chiba Cancer Center, Chiba
  - Kagoshima City Hospital, Kagoshima
  - Kyoto University Hospital, Kyoto
  - Nagasaki University Hospital, Nagasaki
  - Niigata University Medical & Dental Hospital, Niigata

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Itamochi H, Takeshima N, Hamanishi J, Hasegawa K, Matsuura M, Miura K, Nagao S, Nakai H, Tanaka N, Tokunaga H, Nishio S, Watari H, Yokoyama Y, Kase Y, Sumino S, Kato A, Suri A, Yasuoka T, Takehara K. Niraparib in Japanese patients with platinum-sensitive recurrent ovarian cancer: final results of a multicenter phase 2 study. J Gynecol Oncol. 2024 Sep;35(5):e115. doi: 10.3802/jgo.2024.35.e115. Epub 2024 Jul 17. PMID 39058367
- [Derived] Takehara K, Matsumoto T, Hamanishi J, Hasegawa K, Matsuura M, Miura K, Nagao S, Nakai H, Tanaka N, Tokunaga H, Ushijima K, Watari H, Yokoyama Y, Kase Y, Sumino S, Suri A, Itamochi H, Takeshima N. Phase 2 single-arm study on the safety of maintenance niraparib in Japanese patients with platinum-sensitive relapsed ovarian cancer. J Gynecol Oncol. 2021 Mar;32(2):e21. doi: 10.3802/jgo.2021.32.e21. Epub 2021 Jan 6. PMID 33470063
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b60284db2bf003ab49986?idFilter=%5B%22Niraparib-2001%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 27 investigative sites in Japan from 28 December 2018 to 28 December 2022.
Pre-assignment Details: Participants with a diagnosis of with platinum-sensitive, relapsed ovarian cancer, fallopian tube cancer, or primary peritoneal cancer, who had achieved complete response (CR) or partial response (PR) in the last chemotherapy containing platinum-based anticancer agents were enrolled to received niraparib 300 mg in this study.
Period: Overall Study
Arm/Group | Niraparib 300 mg
Started | 19
Response Evaluable Set (Response-evaluable analysis set includes participants who had measurable disease at baseline.) | 5
Completed | 0
Not Completed | 19
Not completed — Adverse Event | 5
Not completed — Progressive Disease | 10
Not completed — Site Terminated by Sponsor | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included participants who received at least 1 dose of study drug.
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (9.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 19
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 19
Height [Mean (Standard Deviation); unit: cm] | 156.7 (4.82)
Weight [Mean (Standard Deviation); unit: kg] | 57.47 (10.445)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index=weight (kg)/[height (m)^2]
  kg/m^2 | 23.46 (4.471)
Breast Cancer (Gene) (BRCA1) Mutant [Count of Participants; unit: Participants] — Participants with mutation of BRCA1 gene.
  Participants
    Without Mutant | 1
    Unknown | 18
BRCA2 Mutant [Count of Participants; unit: Participants] — Participants with mutation of BRCA2 gene.
  Participants
    Without Mutant | 1
    Unknown | 18
Time to Progression after the Penultimate (Next to Last) Platinum Therapy [Count of Participants; unit: Participants] — Participants with time to progression were categorized as 6-12 months and more than 12 months. Time to progression is defined as the time from the date of last administration of platinum therapy to the first documentation of disease progression.
  Participants
    6-12 Months | 5
    More Than 12 Months | 14
Best Response during the Last Platinum Regimen [Count of Participants; unit: Participants] — Best response is based on the investigators assessment.
  Participants
    Complete Response (CR) | 8
    Partial Response (PR) | 11
Time from Last Platinum Therapy to Start of Study Drug (days) [Median (Full Range); unit: days] — Duration in days from the date of last platinum therapy to the date of start of study drug.
  days | 42.0 [14 to 65]
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — The ECOG scale is as follows: Grade 0: Fully active, able to perform all pre-disease activities without restriction; Grade 1: Restricted in physically strenuous activity, ambulatory, able to carry out light work; Grade 2: Ambulatory and capable of all self-care but unable to work. Up and about more than 50% of waking hours; Grade 3: Capable of only limited self-care, confined to bed or chair > 50% of waking hours; Grade 4: Completely disabled. Cannot carry on any self-care. Only categories with participants is reported.
  Participants
    0 | 17
    1 | 2
Primary Tumor Site [Count of Participants; unit: Participants] — Participants with site of tumor are reported.
  Participants
    Ovarian | 10
    Primary Peritoneal | 5
    Fallopian Tube | 4
Duration Since Initial Diagnosis of Primary Cancer [Median (Full Range); unit: years] — Duration since initial diagnosis is defined as the time elapsed since the first diagnosis to the date of enrolment.
  years | 3.35 [1.2 to 19.6]
Cancer Stage at Time of Initial Diagnosis [Count of Participants; unit: Participants] — Cancer stage was determined based on federation of obstetrics and gynecology(FIGO) staging system. Stage I-Only in ovaries, Stage II-Has grown outside ovaries and is growing within pelvis, Stage III-Has spread outside pelvis into abdominal cavity or to lymph nodes(Stage IIIB-cancer growths ≤2cm in size on lining of abdomen(peritoneum) and there might also be cancer in lymph nodes; Stage IIIC-cancer growths >2cm on lining of abdomen(peritoneum) and might also be in lymph nodes), Stage IV-Has spread to other body organs, Unknown-Data could not be collected for the defined stages.
  Participants
    IC | 1
    IIC | 1
    IIIB | 2
    IIIC | 10
    IV | 4
    Unknown | 1
Sites of Metastatic Disease [Count of Participants; unit: Participants] — All sites of metastatic disease are counted. Population: Number analyzed is the number of participants with sites of metastatic disease at baseline.
  Participants
    number analyzed (Participants) | 8
    Ascites or pleural effusion | 1
    Peritoneum | 4
    Lymph Nodes | 1
    Other | 2
Number of Metastatic Sites [Mean (Standard Deviation); unit: metastatic Sites] — Population: Number analyzed is the number of participants with sites of metastatic disease.
  metastatic Sites
    number analyzed (Participants) | 8
    (all) | 1.0 (0.00)
Prior Radiation Therapy [Count of Participants; unit: Participants]
  Had Radiation Therapy | 1
  Had No Radiation Therapy | 18
Prior Surgery/Procedure [Count of Participants; unit: Participants]
  Had Surgery/ Procedure | 19
Prior Chemotherapy [Count of Participants; unit: Participants]
  Had Chemotherapy | 19
Number of Prior Surgery/Procedure for Study Indication [Mean (Standard Deviation); unit: number of surgery] | 2.3 (1.38)
Prior History of Myelosuppression [Count of Participants; unit: Participants]
  Had Myelosuppression | 19
Prior Thrombocytopenia [Count of Participants; unit: Participants] — Thrombocytopenia was defined as decrease in thrombocytes i.e. platelet count in participant. Thrombocytopenia was graded as per the NCI-CTCAE .As per the NCI-CTCAE, Grade 1 scales as Mild; Grade 2 scales as Moderate; Grade 3 scales as severe or medically significant but not immediately life threatening; Grade 4 scales as life-threatening consequences; and Grade 5 scales as death related to Adverse Events (AE). Population: Number analyzed is the number of participants with prior thrombocytopenia at baseline.
  Participants
    number analyzed (Participants) | 18
    Grade 1 | 12
    Grade 2 | 2
    Grade 3 | 3
    Grade 4 | 1
Prior Leukopenia [Count of Participants; unit: Participants] — Leukopenia is defined as decrease in the leukocytes i.e white blood cells in participant. Leukopenia was graded as per the NCI-CTCAE. As per the NCI-CTCAE, Grade 1 scales as Mild; Grade 2 scales as Moderate; Grade 3 scales as severe or medically significant but not immediately life threatening; Grade 4 scales as life-threatening consequences; and Grade 5 scales as death related to Adverse Events (AE). Only categories with participants is reported. Population: Number analyzed is the number of participants with prior leukopenia at baseline.
  Participants
    number analyzed (Participants) | 16
    Grade 2 | 6
    Grade 3 | 9
    Grade 4 | 1
Prior Anemia [Count of Participants; unit: Participants] — Anaemia is defined as a condition in which the number of red blood cells or their oxygen-carrying capacity is insufficient to meet physiologic needs. Anaemia was graded as per the NCI-CTCAE. As per the NCI-CTCAE, Grade 1 scales as Mild; Grade 2 scales as Moderate; Grade 3 scales as severe or medically significant but not immediately life threatening; Grade 4 scales as life-threatening consequences; and Grade 5 scales as death related to Adverse Events (AE). Only categories with participants is reported. Population: Number analyzed is the number of participants with prior anemia at baseline.
  Participants
    number analyzed (Participants) | 17
    Grade 1 | 1
    Grade 2 | 5
    Grade 3 | 11
Prior Neutropenia [Count of Participants; unit: Participants] — Neutropenia is defined as low level of neutrophils i.e. white blood cells in participants. Neutropenia was graded as per the NCI-CTCAE. As per the NCI-CTCAE, Grade 1 scales as Mild; Grade 2 scales as Moderate; Grade 3 scales as severe or medically significant but not immediately life threatening; Grade 4 scales as life-threatening consequences; and Grade 5 scales as death related to Adverse Events (AE). Only categories with participants is reported.
  Participants
    Grade 2 | 1
    Grade 3 | 6
    Grade 4 | 12
Baseline Platelets Count [Mean (Standard Deviation); unit: 10^9 platelets/L] | 214.1 (58.06)
Ovarian Cancer Pathology Histological [Count of Participants; unit: Participants] | 19
Tumor Grade [Count of Participants; unit: Participants] — With regard to tumor grading, conventional FIGO/ gynecologic oncology group (GOG)/ world health organisation (WHO) criteria or two-tier system for grading ovarian serous carcinoma is used; participants with grade 3 tumors in FIGO/GOG/WHO criteria (among grade 1 as well differentiated, grade 2 as moderately differentiated, and grade 3 indicates poorly differentiated) or participants with high-grade tumors in two-tier system (among low-grade or high-grade) are enrolled.
  Participants
    Grade 3 | 5
    Higher Grade | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 3 or 4 Thrombocytopenia Occurring Within 30 Days After Initial Administration of Niraparib
Description: An adverse event of 'thrombocytopenia' was collected and graded as per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.03.As per the NCI-CTCAE, Grade 1 scales as Mild; Grade 2 scales as Moderate; Grade 3 scales as severe or medically significant but not immediately life threatening; Grade 4 scales as life-threatening consequences; and Grade 5 scales as death related to Adverse Events (AE).
Time Frame: Up to 30 days after the first dose
Population: Safety Analysis Set included participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 19
Participants | 6

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An AE is defined as any untoward medical occurrence in a participant who has enrolled in a study; it does not necessarily have a causal relationship with this treatment. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: From the day of signing the informed consent form (ICF) until 30 days after last dose of study drug administration or beginning of subsequent anticancer therapy, whichever comes first (up to 48 months).
Population: Safety Analysis Set included participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 19
Participants | 19

3. Secondary Outcome: Number of Participants With Grade 3 or Higher TEAEs
Description: An AE is defined as any untoward medical occurrence in a participant who has enrolled in a study; it does not necessarily have a causal relationship with this treatment. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug. A severity grade is defined by the NCI-CTCAE Version 4.03. As per NCI-CTCAE, Grade 1 scales as Mild; Grade 2 scales as Moderate; Grade 3 scales as severe or medically significant but not immediately life threatening; Grade 4 scales as life-threatening consequences; and Grade 5 scales as death related to AE.
Time Frame: From the day of signing the ICF until 30 days after last dose of study drug administration or beginning of subsequent anticancer therapy, whichever comes first (up to 48 months).
Population: Safety Analysis Set included participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 19
Participants | 14

4. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An SAE is any AE that results in death, is life-threatening, requires inpatient hospitalization or prolongation of an existing hospitalization, results in significant disability or incapacity, is a congenital anomaly/birth defect or is a medically important event.
Time Frame: as for outcome 3
Population: Safety Analysis Set included participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 19
Participants | 4

5. Secondary Outcome: Number of Participants With TEAEs Leading to Drug Discontinuation
Description: as for outcome 2
Time Frame: as for outcome 3
Population: Safety Analysis Set included participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 19
Participants | 5

6. Secondary Outcome: Number of Participants With TEAEs Leading to Dose Interruption
Description: as for outcome 2
Time Frame: as for outcome 3
Population: Safety Analysis Set included participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 19
Participants | 16

7. Secondary Outcome: Number of Participants With TEAEs Leading to Dose Reduction
Description: as for outcome 2
Time Frame: as for outcome 3
Population: Safety Analysis Set included participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 19
Participants | 16

8. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time in months from the date of first study drug administration to the date of first documentation of progressive disease (PD) or death as assessed by the Investigator per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Per RECIST 1.1, PD is defined as at least a 20% increase in the SoD (Sum of Diameters) of target lesions, taking as a reference the smallest (nadir) SoD since (and including) baseline. In addition to the relative increase of 20%, the SoD must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From first study drug administration until disease progression or death (up to 48 months)
Population: Full Analysis Set included participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: months
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 19
months | 18 [1.8 to 46]

9. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the study enrollment to death due to any cause.
Time Frame: Up to 48 months
Population: Full Analysis Set included participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: months
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 19
months | NA [14.3 to 47] — Median was not estimable due to low number of participants with events.

10. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the proportion of participants achieving Complete Response (CR) or Partial Response (PR) as assessed by the investigator per RECIST (v.1.1). Per RECIST 1.1, CR is defined as disappearance of all target lesions; PR is defined as atleast 30% decrease in sum of diameters (SoD) of target lesions.
Time Frame: Up to 48 months
Population: Response-evaluable Analysis Set included participants who received at least 1 dose of study drug and had at least one measurable disease at baseline. The data is reported only for responders.
Measure: Number; unit: percentage of participants
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 5
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: From the day of signing the ICF until 30 days after last dose of study drug administration or beginning of subsequent anticancer therapy, whichever comes first (up to 48 months).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Niraparib 300mg: Niraparib 300 mg, capsules, orally, once daily on Days 1 to 28 of each 28-day treatment cycle (up to 51 cycles).
Arm/Group | Niraparib 300mg
All-Cause Mortality (participants affected / at risk) | 6/19
Serious Adverse Events (participants affected / at risk) | 4/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Niraparib 300mg (N=19)
Bile duct stone (Hepatobiliary disorders) | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pneumonia (Infections and infestations) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Niraparib 300mg (N=19)
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 4
Alanine aminotransferase increased (Investigations) | 1
Anaemia (Blood and lymphatic system disorders) | 9
Angular cheilitis (Infections and infestations) | 1
Anxiety (Psychiatric disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Aspartate aminotransferase increased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4
Blood creatinine increased (Investigations) | 3
Catheter site thrombosis (General disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Contrast media allergy (Immune system disorders) | 4
Cystitis (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 9
Dehydration (Metabolism and nutrition disorders) | 1
Dental caries (Gastrointestinal disorders) | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 1
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1
Device breakage (Product Issues) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Dizziness (Nervous system disorders) | 1
Dizziness postural (Nervous system disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 2
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1
Head discomfort (Nervous system disorders) | 1
Headache (Nervous system disorders) | 7
Hepatic function abnormal (Hepatobiliary disorders) | 1
Hypertension (Vascular disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Influenza (Infections and infestations) | 1
Infusion site extravasation (General disorders) | 1
Insomnia (Psychiatric disorders) | 2
Intercostal neuralgia (Nervous system disorders) | 1
Laryngitis (Infections and infestations) | 1
Leukopenia (Blood and lymphatic system disorders) | 2
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Malaise (General disorders) | 5
Menopausal symptoms (Reproductive system and breast disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nasopharyngitis (Infections and infestations) | 6
Nausea (Gastrointestinal disorders) | 14
Neuropathy peripheral (Nervous system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 3
Neutrophil count decreased (Investigations) | 11
Occult blood (Investigations) | 1
Oedema peripheral (General disorders) | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 1
Oral herpes (Infections and infestations) | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Palpitations (Cardiac disorders) | 3
Periodontal disease (Gastrointestinal disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Pharyngitis (Infections and infestations) | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1
Platelet count decreased (Investigations) | 12
Pruritus (Skin and subcutaneous tissue disorders) | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Pyrexia (General disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Renal impairment (Renal and urinary disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1
Skin infection (Infections and infestations) | 1
Stomatitis (Gastrointestinal disorders) | 5
Tachycardia (Cardiac disorders) | 1
Thirst (General disorders) | 1
Tinea infection (Infections and infestations) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Vaginal discharge (Reproductive system and breast disorders) | 1
Vomiting (Gastrointestinal disorders) | 9
Vulvitis (Infections and infestations) | 1
Weight decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/87/NCT03759587/Prot_002.pdf
  • Statistical Analysis Plan (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/87/NCT03759587/SAP_001.pdf